CLINICAL TRIAL: NCT04092855
Title: Early Identification and Prediction of Right Ventricular Dysfunction and Failure in Critically Ill Patients: An Observational Non-Interventional Cohort Study
Brief Title: Right Ventricular Pressure Waveform Monitoring in Cardiac Surgery
Acronym: PACEPORT
Status: Recruiting | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Edwards Lifesciences (Industry)
Responsible Party: Principal Investigator, Andre Denault, Principal Investigator, Montreal Heart Institute
Other Study IDs: 2019-2527
Record Dates: First submitted 2019-04-25; First posted 2019-09-17 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Right Ventricular Dysfunction; Right Heart Failure; Congestive Heart Failure
Keywords: Right Ventricular Pressure Waveform
MeSH Terms: conditions — Ventricular Dysfunction, Right; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
RV dysfunction has been associated with increased mortality in the ICU and cardiac surgical patients. Thus, early identification of RV dysfunction at less severe stages will allow for earlier intervention and potentially better patient outcomes.

However, so far, no studies have reported prospectively the prevalence of abnormal RV pressure waveform during cardiac surgery and in the ICU. The investigator's primary hypothesis is that the prevalence of abnormal RV pressure waveform occurs in more than 50% of cardiac surgical patients throughout their hospitalization. Those patients with abnormal RV pressure waveform will be more prone to post-operative complications related to RV dysfunction and failure in the OR and ICU.

DETAILED DESCRIPTION:
Right ventricular (RV) dysfunction is mostly associated to a decrease in contractility, right ventricular pressure overload or right ventricular volume overload. RV dysfunction can occur in a number of clinical scenarios in the intensive care unit (ICU) and operating room (OR): pulmonary embolism, acute respiratory distress syndrome (ARDS), septic shock, RV infarction, and in pulmonary hypertensive patients undergoing cardiac surgery.

Unfortunately, identifying which patients will develop RV dysfunction and then progress towards RV failure have proven difficult. One of the reasons for delaying the diagnosis of RV dysfunction could be the lack of uniform definition, especially in the perioperative period. Echocardiographic definitions of RV dysfunction have been described: RV fractional area change (RVFAC) < 35 %, tricuspid annular plane systolic excursion (TAPSE) < 16 mm, tissue Doppler S wave velocity <10 cm/s, RV ejection fraction (RVEF) <45% and RV dilation. However, echocardiographic indices alone are insufficient in describing RV function. The diagnosis of fulminant RV failure is more easily recognised as a combination of echocardiographic measures, compromised hemodynamic measures and clinical presentation. RV dysfunction is inevitably associated with absolute or relative pulmonary hypertension because of the anatomic and physiological connection between the RV and pulmonary vascular system. The gold standard for measuring pulmonary pressure is still the pulmonary artery catheter. However, RV output can initially be preserved despite of pulmonary hypertension. It is therefore mandatory that early, objective, continuous, easily obtainable and subclinical indices of RV dysfunction are found and validated to initiate early treatment of this disease.

ELIGIBILITY:
Inclusion Criteria:

-Male or female patients, age 18 and older, undergoing cardiac surgery and receiving standard of care monitoring utilizing a pulmonary artery catheter.

Exclusion Criteria:

* Emergency surgery or inability to obtain consent
* Concomitant diseases such as pericardial constriction, congenital heart disease, severe valvular regurgitation, right ventricular systolic dysfunction, or right ventricular infarction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing cardiac surgery.
Sampling Method: Probability Sample
Enrollment: 112 (Estimated)
Dates: Start 2018-12-10 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of abnormal diastolic RV waveforms before CPB, after CPB and in the ICU | From thermodilution catheter insertion until 2 hours after ICU arrival
  Abnormal RV pressure waveform will be defined as a difference between the RV end-diastolic minus the early-diastolic pressure > 4 mmHg.

SECONDARY OUTCOMES:
Proportion of patients with difficult and complex separation from cardiopulmonary bypass at the end of cardiac surgery | From the discontinuation of cardiopulmonary bypass until ICU arrival after surgery, assessed up to 4 hours.
  Difficult separation from cardiopulmonary bypass: instability requiring at least two different types of pharmacological agents (i.e., inotropes ± vasopressors ± inhaled agents) Complex separation from cardiopulmonary bypass: Hemodynamic instability requiring return on cardiopulmonary bypass or addition of mechanical support (intra-aortic balloon pump or extra-corporeal membrane oxygenator)
Cumulative time of Persistent Organ Dysfunction or Death (TPOD) during the first 28 days after cardiac surgery | Up to 28 days or until hospital discharge
  TPOD is a continuous variable representative of the burden of care and morbidity during the first 28 days following cardiac surgery and was chosen to circumvent issues arising for using other clinical endpoint such as ICU length of stay
Incidence of deaths during hospitalisation | Up to 30 days or until hospital discharge
  Death from any cause
Incidence of acute kidney injury (AKI) | Up to 28 days or until hospital discharge
  Acute kidney injury (AKI) according to KDIGO serum creatinine criteria:
  Stage 1: ≥50% or 27 umol/L increases in serum creatinine, Stage 2: ≥100% increase in serum creatinine, Stage 3 ≥200% increase in serum creatinine or an increase to a level of ≥254 umol/L or dialysis initiation.
Incidence of major bleeding | Up to 28 days or until hospital discharge
  Major bleeding is defined by the Bleeding Academic Research Consortium (BARC) as one of the following:
  * Perioperative intracranial bleeding within 48h
  * Reoperation after closure of sternotomy for the purpose of controlling bleeding
  * Transfusion of ≥5 units of whole blood of packed red blood cells within a 48 hours period
  * Chest tube output ≥2L within a 24 hours period
Incidence of surgical reintervention for any reasons | Up to 28 days or until hospital discharge
  Re-operation after the initial surgery for any cause
Incidence of deep sternal wound infection or mediastinitis | Up to 28 days or until hospital discharge
  Diagnosis of a deep incisional surgical site infection or mediastinitis by a surgeon or attending physician
Incidence of delirium | Up to 28 days or until hospital discharge
  Delirium is defined as an intensive care delirium screening checklist (ICDSC) score(18) of ≥4 in the week following surgery or positive result for the Confusion Assessment Method for the ICU (CAM-ICU).
Incidence of stroke | Up to 28 days or until hospital discharge
  Central neurologic deficit persisting longer than 72 hours
Total duration of ICU stay in hours | Up to 28 days or until hospital discharge
  Number of hours passed in the ICU
Duration of vasopressor requirements (in hours) | Up to 28 days or until hospital discharge
  Vasopressors include norepinephrine, epinephrine, dobutamine, vasopressin, phenylephrine, milrinone, isoproterenol and dopamine.
Duration of hospital stay (in days) | Up to 28 days or until hospital discharge
  Number of days hospitalized from the day of surgery to discharge
Duration of mechanical ventilation (in hours) | Up to 28 days or until hospital discharge
  A duration of >24 hours will be considered prolonged ventilation requirements.
Incidence of major morbidity or mortality | Up to 28 days or until hospital discharge
  Including death, prolonged ventilation, stroke, renal failure (Stage ≥2), deep sternal wound infection and reoperation for any reason.
Right ventricular ejection fraction | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Right ventricular fractional area change | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Right ventricular strain | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Tricuspid annular plane systolic excursion | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Right ventricular performance index | From arrival to the operating room until 2 hours after ICU arrival
  Assessed by the American Society of Echocardiography guidelines
Portal flow pulsatility fraction | From arrival to the operating room until 2 hours after ICU arrival
  Defined as the difference between the maximal and the minimal velocity during the cardiac cycle divided by the maximal velocity
Right ventricular stroke work index | From arrival to the operating room until 2 hours after ICU arrival
  0.0136x Stroke volume index x (Mean pulmonary artery pressure-mean right atrial pressure)
Relative pulmonary pressure | From arrival to the operating room until 2 hours after ICU arrival
  The ratio of the mean systemic arterial pressure divided by the mean pulmonary artery pressure
Right ventricular function index | From arrival to the operating room until 2 hours after ICU arrival
  Defined as (isovolumic contraction time + isovolumic relaxation time)/RV ejection time
Pulmonary artery pulsatility index (PAPi) | From arrival to the operating room until 2 hours after ICU arrival
  Defined as (systolic pulmonary artery pressure - diastolic pulmonary artery pressure)/central venous pressure]
Compliance of the pulmonary artery (CPA) | From arrival to the operating room until 2 hours after ICU arrival
  Stroke volume divided by the pulmonary artery pulse pressure (systolic minus the diastolic pulmonary artery pressure)
Pulsatility of femoral venous flow | From arrival to the operating room until 2 hours after ICU arrival
  Velocity variations of blood flow in the femoral vein during the cardiac cycle

CONTACTS AND LOCATIONS:
Overall Officials: Andre Denault, MD,PhD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Haddad F, Doyle R, Murphy DJ, Hunt SA. Right ventricular function in cardiovascular disease, part II: pathophysiology, clinical importance, and management of right ventricular failure. Circulation. 2008 Apr 1;117(13):1717-31. doi: 10.1161/CIRCULATIONAHA.107.653584. No abstract available. PMID 18378625
- [Background] Denault AY, Bussières J, Carrier M, Mathieu P, and the DSBSG. The importance of difficult separation from cardiopulmonary bypass: the Montreal and Quebec Heart Institute experience. Exp Clin Cardiol. 2006;11 (1):37.
- [Background] Denault AY, Bussieres JS, Arellano R, Finegan B, Gavra P, Haddad F, Nguyen AQN, Varin F, Fortier A, Levesque S, Shi Y, Elmi-Sarabi M, Tardif JC, Perrault LP, Lambert J. A multicentre randomized-controlled trial of inhaled milrinone in high-risk cardiac surgical patients. Can J Anaesth. 2016 Oct;63(10):1140-1153. doi: 10.1007/s12630-016-0709-8. Epub 2016 Jul 28. PMID 27470232
- [Background] Rudski LG, Lai WW, Afilalo J, Hua L, Handschumacher MD, Chandrasekaran K, Solomon SD, Louie EK, Schiller NB. Guidelines for the echocardiographic assessment of the right heart in adults: a report from the American Society of Echocardiography endorsed by the European Association of Echocardiography, a registered branch of the European Society of Cardiology, and the Canadian Society of Echocardiography. J Am Soc Echocardiogr. 2010 Jul;23(7):685-713; quiz 786-8. doi: 10.1016/j.echo.2010.05.010. No abstract available. PMID 20620859
- [Background] Raymond M, Gronlykke L, Couture EJ, Desjardins G, Cogan J, Cloutier J, Lamarche Y, L'Allier PL, Ravn HB, Couture P, Deschamps A, Chamberland ME, Ayoub C, Lebon JS, Julien M, Taillefer J, Rochon A, Denault AY. Perioperative Right Ventricular Pressure Monitoring in Cardiac Surgery. J Cardiothorac Vasc Anesth. 2019 Apr;33(4):1090-1104. doi: 10.1053/j.jvca.2018.08.198. Epub 2018 Aug 25. PMID 30269893
- [Background] Haddad F, Couture P, Tousignant C, Denault AY. The right ventricle in cardiac surgery, a perioperative perspective: I. Anatomy, physiology, and assessment. Anesth Analg. 2009 Feb;108(2):407-21. doi: 10.1213/ane.0b013e31818f8623. PMID 19151264
- [Background] Naeije R, Manes A. The right ventricle in pulmonary arterial hypertension. Eur Respir Rev. 2014 Dec;23(134):476-87. doi: 10.1183/09059180.00007414. PMID 25445946
- [Background] Denault AY, Chaput M, Couture P, Hebert Y, Haddad F, Tardif JC. Dynamic right ventricular outflow tract obstruction in cardiac surgery. J Thorac Cardiovasc Surg. 2006 Jul;132(1):43-9. doi: 10.1016/j.jtcvs.2006.03.014. PMID 16798301
- [Background] Denault A, Lamarche Y, Rochon A, Cogan J, Liszkowski M, Lebon JS, Ayoub C, Taillefer J, Blain R, Viens C, Couture P, Deschamps A. Innovative approaches in the perioperative care of the cardiac surgical patient in the operating room and intensive care unit. Can J Cardiol. 2014 Dec;30(12 Suppl):S459-77. doi: 10.1016/j.cjca.2014.09.029. Epub 2014 Oct 5. PMID 25432139
- [Background] St-Pierre P, Deschamps A, Cartier R, Basmadjian AJ, Denault AY. Inhaled milrinone and epoprostenol in a patient with severe pulmonary hypertension, right ventricular failure, and reduced baseline brain saturation value from a left atrial myxoma. J Cardiothorac Vasc Anesth. 2014 Jun;28(3):723-9. doi: 10.1053/j.jvca.2012.10.017. Epub 2013 Apr 26. No abstract available. PMID 23623891
- [Background] Amsallem M, Kuznetsova T, Hanneman K, Denault A, Haddad F. Right heart imaging in patients with heart failure: a tale of two ventricles. Curr Opin Cardiol. 2016 Sep;31(5):469-82. doi: 10.1097/HCO.0000000000000315. PMID 27467173
- [Background] Korshin A, Gronlykke L, Nilsson JC, Moller-Sorensen H, Ihlemann N, Kjoller M, Damgaard S, Lehnert P, Hassager C, Kjaergaard J, Ravn HB. The feasibility of tricuspid annular plane systolic excursion performed by transesophageal echocardiography throughout heart surgery and its interchangeability with transthoracic echocardiography. Int J Cardiovasc Imaging. 2018 Jul;34(7):1017-1028. doi: 10.1007/s10554-018-1306-4. Epub 2018 Jan 30. PMID 29383465
- [Background] Hrymak C, Strumpher J, Jacobsohn E. Acute Right Ventricle Failure in the Intensive Care Unit: Assessment and Management. Can J Cardiol. 2017 Jan;33(1):61-71. doi: 10.1016/j.cjca.2016.10.030. Epub 2016 Nov 11. PMID 28024557
- [Background] Stoppe C, McDonald B, Benstoem C, Elke G, Meybohm P, Whitlock R, Fremes S, Fowler R, Lamarche Y, Jiang X, Day AG, Heyland DK. Evaluation of Persistent Organ Dysfunction Plus Death As a Novel Composite Outcome in Cardiac Surgical Patients. J Cardiothorac Vasc Anesth. 2016 Jan;30(1):30-8. doi: 10.1053/j.jvca.2015.07.035. Epub 2015 Jul 29. PMID 26847748
- [Background] Rubenfeld GD, Angus DC, Pinsky MR, Curtis JR, Connors AF Jr, Bernard GR. Outcomes research in critical care: results of the American Thoracic Society Critical Care Assembly Workshop on Outcomes Research. The Members of the Outcomes Research Workshop. Am J Respir Crit Care Med. 1999 Jul;160(1):358-67. doi: 10.1164/ajrccm.160.1.9807118. No abstract available. PMID 10390426
- [Background] Kellum JA, Lameire N; KDIGO AKI Guideline Work Group. Diagnosis, evaluation, and management of acute kidney injury: a KDIGO summary (Part 1). Crit Care. 2013 Feb 4;17(1):204. doi: 10.1186/cc11454. PMID 23394211
- [Background] Mehran R, Rao SV, Bhatt DL, Gibson CM, Caixeta A, Eikelboom J, Kaul S, Wiviott SD, Menon V, Nikolsky E, Serebruany V, Valgimigli M, Vranckx P, Taggart D, Sabik JF, Cutlip DE, Krucoff MW, Ohman EM, Steg PG, White H. Standardized bleeding definitions for cardiovascular clinical trials: a consensus report from the Bleeding Academic Research Consortium. Circulation. 2011 Jun 14;123(23):2736-47. doi: 10.1161/CIRCULATIONAHA.110.009449. No abstract available. PMID 21670242
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Inouye SK, van Dyck CH, Alessi CA, Balkin S, Siegal AP, Horwitz RI. Clarifying confusion: the confusion assessment method. A new method for detection of delirium. Ann Intern Med. 1990 Dec 15;113(12):941-8. doi: 10.7326/0003-4819-113-12-941. PMID 2240918
- [Background] Sun LY, Chung AM, Farkouh ME, van Diepen S, Weinberger J, Bourke M, Ruel M. Defining an Intraoperative Hypotension Threshold in Association with Stroke in Cardiac Surgery. Anesthesiology. 2018 Sep;129(3):440-447. doi: 10.1097/ALN.0000000000002298. PMID 29889106
- [Background] Shahian DM, O'Brien SM, Filardo G, Ferraris VA, Haan CK, Rich JB, Normand SL, DeLong ER, Shewan CM, Dokholyan RS, Peterson ED, Edwards FH, Anderson RP; Society of Thoracic Surgeons Quality Measurement Task Force. The Society of Thoracic Surgeons 2008 cardiac surgery risk models: part 1--coronary artery bypass grafting surgery. Ann Thorac Surg. 2009 Jul;88(1 Suppl):S2-22. doi: 10.1016/j.athoracsur.2009.05.053. PMID 19559822
- [Background] Denault AY, Pearl RG, Michler RE, Rao V, Tsui SS, Seitelberger R, Cromie M, Lindberg E, D'Armini AM. Tezosentan and right ventricular failure in patients with pulmonary hypertension undergoing cardiac surgery: the TACTICS trial. J Cardiothorac Vasc Anesth. 2013 Dec;27(6):1212-7. doi: 10.1053/j.jvca.2013.01.023. Epub 2013 Mar 21. PMID 23523254
- [Background] Ait-Oufella H, Bourcier S, Alves M, Galbois A, Baudel JL, Margetis D, Bige N, Offenstadt G, Maury E, Guidet B. Alteration of skin perfusion in mottling area during septic shock. Ann Intensive Care. 2013 Sep 16;3(1):31. doi: 10.1186/2110-5820-3-31. PMID 24040941
- [Background] Vieillard-Baron A, Naeije R, Haddad F, Bogaard HJ, Bull TM, Fletcher N, Lahm T, Magder S, Orde S, Schmidt G, Pinsky MR. Diagnostic workup, etiologies and management of acute right ventricle failure : A state-of-the-art paper. Intensive Care Med. 2018 Jun;44(6):774-790. doi: 10.1007/s00134-018-5172-2. Epub 2018 May 9. PMID 29744563
- [Background] Beaubien-Souligny W, Benkreira A, Robillard P, Bouabdallaoui N, Chasse M, Desjardins G, Lamarche Y, White M, Bouchard J, Denault A. Alterations in Portal Vein Flow and Intrarenal Venous Flow Are Associated With Acute Kidney Injury After Cardiac Surgery: A Prospective Observational Cohort Study. J Am Heart Assoc. 2018 Oct 2;7(19):e009961. doi: 10.1161/JAHA.118.009961. PMID 30371304
- [Derived] Hammoud A, Mailhot T, Parent M, Huard K, Lachance O, Tawil P, Calderone A, Levesque S, Jarry S, Beaubien-Souligny W, Couture EJ, Denault AY. Femoral Vein Pulsatility and Neurocognitive Disorder in Cardiac Surgery. CJC Open. 2024 Nov 8;7(2):187-192. doi: 10.1016/j.cjco.2024.11.002. eCollection 2025 Feb. PMID 40060204